CLINICAL TRIAL: NCT01516047
Title: An Open-Label Pharmacokinetic Study of Abiraterone Acetate Suspension in Subjects With Severe Hepatic Impairment Compared to Matched Control Subjects With Normal Hepatic Function
Brief Title: A Pharmacokinetic Study of Abiraterone Acetate in Patients With Severe Hepatic Impairment Compared to Patients With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100779; 212082PCR1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Pharmacology; Pharmacokinetics; Pharmacodynamics; Abiraterone acetate suspension; JNJ-212082
MeSH Terms: interventions — KPNA1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Patients with severe hepatic impairment.
  Interventions: Drug: Cohort 1
- Cohort 2 (Experimental): Healthy individuals with normal hepatic function.
  Interventions: Drug: Cohort 2

INTERVENTIONS:
Drug: Cohort 1 — 125 mg to 2000 mg abiraterone acetate suspension on Day 1
  Arms: Cohort 1
Drug: Cohort 2 — 2000 mg abiraterone acetate suspension on Day 1
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to evaluate systemic exposure of abiraterone acetate in adult male patients with severe hepatic impairment and is being conducted to collect information that will support clinical dosing recommendations for this subpopulation.

DETAILED DESCRIPTION:
This is a non-randomized (individuals will not be assigned by chance to study treatments), open-label (individuals will know the identity of study treatments), single dose, 2-cohort study of abiraterone acetate in approximately 16 adult men. Participants will either have severe hepatic impairment (Cohort 1) or qualify for the control group with normal hepatic function (Cohort 2). This study will consist of a screening period followed by a 4-day open-label treatment phase and subsequently a 28-day follow up after the study dose of abiraterone acetate suspension. Patients will be admitted to the study center on Day -1, a single dose of study drug will be administered on the morning of Day 1, and patients will remain at the study center until completion of the 72-hour pharmacokinetic (PK; study of what the body does to a drug) blood sample collection in the morning of Day 4. Enrollment will begin sequentially with patients in the severe hepatic impairment cohort. Enrollment for Cohort 1 will be staggered in order to evaluate safety and tolerability. The study will not proceed if >=Grade 3 toxicity or serious adverse events considered related to abiraterone acetate are observed. Additional patients may be enrolled if at least 8 patients in each cohort do not complete the required assessments, including the PK blood sample collections. The aim will be to treat the remaining patients in Cohort 1 at a suspension dose yielding an exposure equivalent to 1000 mg tablet in healthy individuals. If the dose is adjusted after Study Evaluation Team review, additional patients may be enrolled to ensure at least 8 patients complete the study at the final dose. Once enrollment of patients in the severe hepatic impairment cohort is completed, the matched-control cohort will be dosed. Serial PK samples will be collected during the open-label treatment phase as detailed in the protocol. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* All participants are to be cancer free and have a body mass index (BMI) between 18 kg/m2 to 40 kg/m2, inclusive, and body weight not less than 50 kg.
* Cohort 1is characterized by severe hepatic impairment (as described by the Child-Pugh Classification C).
* Cohort 2 represents a matched control characterized by healthy participants with normal hepatic function.
* Control cohort participants will be age matched ± 10 years and BMI matched within 20% of the means of the severe hepatic impairment cohort; no other clinical criteria will be matched.
* Control cohort participants must be in good health, with no clinically significant findings from medical history, physical examination, laboratory evaluations, 12-lead electrocardiogram and vital signs.
* Patients with hepatic impairment are required to be on medication and/or treatment regimen to treat their underlying hepatic impairment or medical conditions before dosing with study drug.

Exclusion Criteria:

* Participants in the control cohort who test positive for hepatitis B surface antigen (HBsAg) or hepatitis C antibodies will not be permitted to enroll in the study.
* Patients with hepatic impairment who have acute or exacerbating hepatitis, fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment in the judgment of either the investigator or the sponsor's medical monitor will be excluded from participating in the study.
* Patients with hepatic impairment taking antiviral therapy for treatment of active hepatitis infection at the time of screening, previously diagnosed with hepatocellular carcinoma, or who have a history of biliary sepsis within the past 2 years.
* Patients with severe hepatic impairment should not have Gilbert's syndrome or >= Grade 3 hepatic encephalopathy where the patient lacks the capacity to provide informed consent as judged by the investigator. Mild or moderate hepatic encephalopathy that would not impede informed consent in the investigator's judgment is permitted.

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Mean plasma concentrations of abiraterone | Up to Day 4
Mean plasma protein binding concentrations of abiraterone | Screening Day -2
Maximum plasma concentrations of abiraterone | Up to Day 4
Time to reach the maximum plasma concentration of abiraterone | Up to Day 4
Area under the plasma concentration-time curve from time 0 to 24 hours after dosing of abiraterone | Up to Day 4
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration of abiraterone | Up to Day 4
Area under the plasma concentration-time curve from time 0 to infinite time of abiraterone | Up to Day 4
Percentage of area under the plasma concentration-time curve from time 0 to infinite time obtained by extrapolation of abiraterone | Up to Day 4
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of abiraterone | Up to Day 4
Time to last quantifiable plasma concentration of abiraterone | Up to Day 4
Total apparent clearance of drug after extravascular administration uncorrected for absolute bioavailability of abiraterone | Up to Day 4
Apparent volume of distribution after extravascular administration uncorrected for absolute bioavailability of abiraterone | Up to Day 4

SECONDARY OUTCOMES:
The number of participants affected by an adverse event | Up to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Research, Study Director — Janssen Research & Development, LLC
Locations (3):
- United States (3):
  - Anaheim, California
  - Orlando, Florida
  - San Antonio, Texas

REFERENCES:
- [Derived] Marbury T, Lawitz E, Stonerock R, Gonzalez M, Jiao J, Breeding J, Haqq C, Verboven P, Stieltjes H, Yu M, Molina A, Acharya M, Chien C, Tran N. Single-dose pharmacokinetic studies of abiraterone acetate in men with hepatic or renal impairment. J Clin Pharmacol. 2014 Jul;54(7):732-41. doi: 10.1002/jcph.253. Epub 2014 Jan 17. PMID 24374856
- See also: An Open-Label Pharmacokinetic Study of Abiraterone Acetate Suspension in Subjects with Severe Hepatic Impairment Compared to Matched Control Subjects with Normal Hepatic Function — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3447&filename=CR100779_CSR.pdf